CLINICAL TRIAL: NCT00570830
Title: Combined Fluocinolone Acetonide Sustained Drug Delivery System Implantation and Phacoemulsification/Intraocular Lens Implantation in Patients With Severe Uveitis
Brief Title: Retisert and Cataract Surgery in Patients With Severe Uveitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Glenn J Jaffe, MD, Duke University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9145; 9145-06--10R0ER
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2008-08

CONDITIONS: Intermediate Uveitis; Posterior Uveitis
MeSH Terms: conditions — Uveitis, Intermediate; Uveitis, Posterior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): single armed case series in which all patients underwent the same treatment.
  Interventions: Device: Retisert (fluocinolone acetonide implant)

INTERVENTIONS:
Device: Retisert (fluocinolone acetonide implant) — Patients with intermediate, posterior or pan-uveitis underwent simultaneous fluocinolone acetonide implantation (0.59 mg or 2.1 mg) and phacoemulsification and intraocular lens.
  Other Names: 1

SUMMARY:
To review chart data at the Duke Eye Center and determined whether a 3-year fluocinolone acetonide sustained drug delivery system (FA) safely suppressed postoperative inflammation when combined with phacoemulsification and posterior chamber intraocular lens implantation (phaco/PCIOL) in eyes with severe uveitis.

DETAILED DESCRIPTION:
Cataracts are common in eyes with uveitis. It results from inflammation or the use of topical or systemic steroids. Cataract surgery can cause an unusually severe inflammatory response, abnormal or excessive bleeding, and unexpected postoperative IOP responses such as hypertension or hypotony. Previous studies showed that successful outcome is preoperative and postoperative control of intraocular inflammation by topical, periocular, and systemic steroidal or immunosuppressive agents. In patients with severe posterior uveitis, periocular and intravitreal injections often provide only transient effects and are associated with complications such as hemorrhage, retinal detachment and endophthalmitis. Oral corticosteroid therapy are also associated with side effects to multiple organ systems in the body. A novel technology that delivers corticosteroid therapy linearly via an intravitreal, polymer-coated, sustained release implant has been developed and FDA approved to treat severe posterior segment uveitis. FA implantation effectively controls inflammation over an extended period of time in a complicated group of patients with posterior and/or panuveitis and allows reduced immunosuppression. We hope to determined whether this implant, a fluocinolone acetonide sustained drug delivery system (FA), can safely suppress postoperative inflammation when combined with phacoemulsification and posterior chamber intraocular lens implantation (phaco/PCIOL) in eyes with severe uveitis. We hypothesize that combining the implant with cataract surgery will provide better surgical outcomes by suppressing inflammation during the postoperative period. By reviewing our own surgical data at the Duke Eye Center, we intend to primarily focus on the safety and effectiveness of this surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* A visually significant cataract
* A history of recurrent noninfectious posterior uveitis or intermediate uveitis with or without iridocyclitis
* incomplete therapeutic response or treatment-limiting side effects to oral, periocular corticosteroid, and/or immunosuppressive agents
* VA of at least light perception; and
* Ability to comprehend informed consent and comply with follow-up examinations

Exclusion Criteria:

* An allergy to fluocinolone acetonide or any component of the delivery system
* A toxoplasmosis scar was present in the study eye,
* A peripheral retinal detachment (RD) in the area of the planned fluocinolone acetonide implant placement
* Required chronic systemic corticosteroid therapy or systemic immunosuppressive therapy to treat non-ocular disease or if they tested positive for human immunodeficiency virus.
* Also excluded were female patients who were pregnant or lactating or not taking precautions to avoid pregnancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-09; Primary Completion 2007-11 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Preoperative and postoperative ocular inflammation | up to 12 months postoperatively

SECONDARY OUTCOMES:
visual acuity | up to 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J Jaffe, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Foster CS, Fong LP, Singh G. Cataract surgery and intraocular lens implantation in patients with uveitis. Ophthalmology. 1989 Mar;96(3):281-8. doi: 10.1016/s0161-6420(89)32898-3. PMID 2629713
- [Background] Jaffe GJ, Martin D, Callanan D, Pearson PA, Levy B, Comstock T; Fluocinolone Acetonide Uveitis Study Group. Fluocinolone acetonide implant (Retisert) for noninfectious posterior uveitis: thirty-four-week results of a multicenter randomized clinical study. Ophthalmology. 2006 Jun;113(6):1020-7. doi: 10.1016/j.ophtha.2006.02.021. Epub 2006 May 9. PMID 16690128
- [Derived] Chieh JJ, Carlson AN, Jaffe GJ. Combined fluocinolone acetonide intraocular delivery system insertion, phacoemulsification, and intraocular lens implantation for severe uveitis. Am J Ophthalmol. 2008 Oct;146(4):589-594. doi: 10.1016/j.ajo.2008.05.035. Epub 2008 Jul 17. PMID 18639220